CLINICAL TRIAL: NCT04812197
Title: A Single Cohort Study to Characterize Differences in Microbial Diversity Between Inflamed and Non-Inflamed Skin of Patients With Immune Checkpoint Inhibitor-Induced Dermatitis
Brief Title: Microbial Diversity Between Inflamed and Non-inflamed Skin of Patients With Immune Checkpoint Inhibitor-Induced Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20378; NCI-2021-00221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20378 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Genito-Urinary Neoplasm
MeSH Terms: conditions — Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Skin Biopsies (Other): Patients undergo punch biopsies of inflamed and non-inflamed skin and a blood sample collection.
  Interventions: Procedure: Biospecimen Collection(Punch Biopsy)

INTERVENTIONS:
Procedure: Biospecimen Collection(Punch Biopsy) — Punch Biopsy of Skin
  Other Names: Biospecimen Collection (Punch Biopsy)

SUMMARY:
This study determines microbial diversity between inflamed and non-inflamed skin of patients with immune checkpoint inhibitor-induced dermatitis. Skin has millions of bacteria. When treated with an immunotherapy agent, skin issues like a rash are common, occurring in up to 45% of patients. This study finds out if the type of bacteria on skin is different between the affected and unaffected skin in patients who have this treatment-related rash and also compares the immune cells found in the skin tissue to those seen in the blood.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if skin microbial diversity (estimated by the Shannon Index) significantly differs between inflamed and non-inflamed skin from patients who have immune checkpoint inhibitor (ICI)-induced dermatitis.

SECONDARY OBJECTIVES:

I. To investigate if certain bacterial species and strains are present in higher concentrations of inflamed versus non-inflamed skin of patients with ICI-induced dermatitis.

II. To compare the immune cell phenotypes of inflamed and non-inflamed skin from patients who have ICI-induced dermatitis.

III. To characterize the immune cell phenotype in the peripheral blood in patients who have ICI-induced dermatitis.

IV. To elucidate any association between the skin microbial diversity and response to immunotherapy, characterized by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (e.g., durable complete response [CR] versus partial response [PR] versus stable disease [SD] versus primary progressive disease).

V. To ascertain if higher concentrations of certain bacterial species are associated with a response to immunotherapy, characterized by both RECIST and immune response criteria.

VI. To evaluate associations between the non-inflamed skin flora and cancer subtypes (e.g., renal cell carcinoma, bladder cancer, lung cancer).

VII. To examine if skin microbiome is associated with specific demographic characteristics such as age and gender.

OUTLINE:

Patients undergo punch biopsies of inflamed and non-inflamed skin and a blood sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving treatment with any of the Food and Drug Administration (FDA) approved monoclonal antibodies that block CTLA-4, PD-1, PD-L1, or any combination thereof
* Patients recommended to undergo skin biopsy due to a clinical diagnosis of ICI-induced dermatitis as part of routine and standard clinical care are eligible
* Patients must be age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Measurable disease as per RECIST 1.1
* Patients must be able to personally sign and date informed consent indicating that the patient has been informed of all pertinent aspects of the study are eligible

Exclusion Criteria:

* Patients taking antibiotics or who plan to begin taking antibiotics
* Use of topical or systemic steroids within the past 14 days. Inhaled steroids are permitted
* Known medical condition (e.g. a disease associated with chronic skin inflammation such as atopic dermatitis or psoriasis) that, in the investigator's opinion, would increase the risk associated with study participation or interfere with the interpretation of results
* Not recovered to non-dermatologic =< grade 1 toxicities related to any prior therapy
* Pregnant woman will not be enrolled in this study. It is a regulatory requirement that for studies that carry no prospect of benefit to the woman, the research can only enroll pregnant women if the resulting knowledge cannot be obtained by any other means. In this study, there is no prospect of direct benefit to the pregnant women
* Patients with human immunodeficiency virus (HIV), hepatitis B, or C will be excluded from this study
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Association between skin microbial diversity and immune checkpoint inhibitor (ICI)-induced dermatitis | Up to 1 year
  Microbial diversity will be estimated by the Shannon Index.

OTHER OUTCOMES:
Skin microbial diversity | Up to 1 year
  Will be associated with response to therapy. The non-flamed skin of responders versus non-responders will be compared against change in Shannon Index. Both parametric and non-parametric tests will be performed on the data as well as its log-transformation.
Abundances of certain skin bacteria in lesion | Up to 1 year
  Will be associated with a higher rate of dermatologic toxicity with ICI. Similar to the evaluation of microbial diversity, will evaluate the concentrations of specific bacteria of inflamed as compared to non-inflamed skin of a similar phenotype (e.g. sebaceous, moist, or dry). This will entail both an individual bacteria abundance evaluation and clustering analysis.
Specific skin bacteria | Up to 1 year
  Will be associated with higher response to ICI. Will evaluate specific bacteriomic differences between the responders and non-responders via individual bacteria abundance assessment and clustering analysis. Response will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and assessed at the time of each skin biopsy. This will entail both an individual bacteria abundance evaluation and clustering analysis.
Tissue and peripheral immune cell phenotypes of ICI-induced dermatitis (I) | Up to 1 year
  Will use immunohistochemistry to aid in characterizing the dermatologic microenvironment as follows:
  will use immunohistochemistry to aid in characterizing the dermatologic microenvironment. The Human Cytokine 30-plex protein assay (Invitrogen) will be used to characterize the plasma levels of cytokines in pg/mL.
Tissue and peripheral immune cell phenotypes of ICI-induced dermatitis (II) | Up to 1 year
  Will use immunohistochemistry to aid in characterizing the dermatologic microenvironment as follows:
  will use immunohistochemistry to aid in characterizing the dermatologic microenvironment. Fluorochrome-labeled antibodies will be used to characterize the number of myeloid cells.
Tissue and peripheral immune cell phenotypes of ICI-induced dermatitis (III) | Up to 1 year
  Will use immunohistochemistry to aid in characterizing the dermatologic microenvironment as follows:
  will use immunohistochemistry to aid in characterizing the dermatologic microenvironment. EasySep PE-selection kit will be used to characterize the number of T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States